CLINICAL TRIAL: NCT07161297
Title: Remimazolam for Colonoscopy in IBD Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBD-REMI 2223386_1
Record Dates: First submitted 2025-07-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: IBD (Inflammatory Bowel Disease)
Keywords: Inflammatory bowel disease (IBD); Remimazolam; Midazolam
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Participants were assigned to sedation with either remimazolam or midazolam based on a pragmatic, time-based allocation schedule (i.e., all procedures during a given week used the same sedation regimen). This approach was chosen to ensure feasibility and avoid operator or patient selection bias. No individual-level randomization was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 2 (Remimazolam + Fentanyl) (Active Comparator): ARM 2: Participants receive intravenous remimazolam plus fentanyl for procedural sedation during colonoscopy
  Interventions: Drug: Intravenous remimazolam (5 mg initially, with optional 2.5 mg boluses) plus fentanyl (100 mcg) for procedural sedation.
- Arm 1 (Midazolam + Fentanyl) (Active Comparator): Arm Description: ARM 1: Participants receive intravenous midazolam plus fentanyl for procedural sedation during colonoscopy.
  Interventions: Drug: Intravenous midazolam (3 mg initially, with optional 3 mg boluses) plus fentanyl (100 mcg) for procedural sedation.

INTERVENTIONS:
Drug: Intravenous remimazolam (5 mg initially, with optional 2.5 mg boluses) plus fentanyl (100 mcg) for procedural sedation. — - Remimazolam + Fentanyl IV fentanyl 100 mcg is given first, followed after 1 minute by IV remimazolam 5 mg over 1 minute. Additional 2.5 mg boluses may be given every 2 minutes as needed. Colonoscopy starts 1 minute after sedation. Vital signs are monitored throughout.
  Arms: Arm 2 (Remimazolam + Fentanyl)
Drug: Intravenous midazolam (3 mg initially, with optional 3 mg boluses) plus fentanyl (100 mcg) for procedural sedation. — - Midazolam + Fentanyl (≤1000 caratteri) IV fentanyl 100 mcg is given first, followed after 1 minute by IV midazolam 3 mg over 1 minute. Additional midazolam may be administered based on clinical judgment. Colonoscopy starts 1 minute after sedation. Vital signs are monitored throughout.
  Arms: Arm 1 (Midazolam + Fentanyl)

SUMMARY:
The goal of this clinical trial is to compare two sedation regimens-remimazolam and midazolam-for colonoscopy in adult patients with inflammatory bowel disease (IBD), including Crohn's disease and ulcerative colitis.

The main questions it aims to answer are:

* Does remimazolam provide patient satisfaction that is non-inferior to midazolam during colonoscopy?
* Does remimazolam allow faster recovery and discharge readiness compared to midazolam?

Researchers will compare sedation with remimazolam plus fentanyl to sedation with midazolam plus fentanyl to see if remimazolam improves patient experience and procedural efficiency.

Participants will:

* Receive either remimazolam or midazolam, each combined with fentanyl, during their scheduled colonoscopy
* Complete a short questionnaire to rate their satisfaction after the procedure
* Be assessed for recovery using a standardized discharge score at 10 and 20 minutes after the procedure

ELIGIBILITY:
* Inclusion Criteria

  * Age ≥18 years
  * Diagnosis of IBD (CD or UC) for ≥6 months
  * Scheduled colonoscopy for clinical or surveillance purposes
  * Ability to provide informed consent
* Exclusion Criteria

  * ASA class IV
  * Allergy to benzodiazepines, opioids, flumazenil, or naloxone
  * Severe COPD
  * Obstructive sleep apnea
  * BMI >35
  * Pregnancy or lactation
  * Prior multiple ileocolonic resections or subtotal colectomy
  * Inability to complete questionnaires

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-07 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | Immediately post-procedure
  Proportion of patients reporting at least "satisfied" with sedation (Likert scale 1-4, 3 or 4 points)

SECONDARY OUTCOMES:
Patient high satisfaction | Immediately post-procedure
  Proportion reporting "very satisfied" (Likert scale 1-4, 4 points)
Incidence of treatment-emergent adverse events | Throughout the observation period (i.e., until discharge)
  Proportion of patients experiencing any of the following adverse events (occurring after the administration of the study drug):
  * Desaturation: peripheral oxygen saturation (SpO₂) below 90%
  * Tachycardia: heart rate greater than 100 bpm
  * Bradycardia: heart rate less than 50 bpm
  * Hypotension: systolic blood pressure below 90 mmHg
Discharge readiness 10' | 10 minutes post-procedure
  Proportion of patients ready for discharge (PADSS ≥9)
Dischatge readiness 20' | 20 minutes post-procedure
  Proportion of patients ready for discharge (PADSS ≥9)
Maximum net benefit | 10 minutes post-procedure
  Proportion of patients reportinng "very satisfied" with sedation (Likert scale 1-4, 4 points) + ready for discharge (PADSS ≥9)

OTHER OUTCOMES:
Endoscopy metrics - cecal intubation rate | During procedure
  Percentage of procedures where the endoscope successfully reaches the cecum and can be visually confirmed by inspecting the appendiceal orifice
Endoscopy metrics - cecal intubation time | During procedure
  Time from the insertion of the colonoscope tip into the anal verge until reaching the cecal base

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes may be shared with qualified researchers upon reasonable request and subject to institutional and ethical approval. Data will be available after publication and will include demographic data, sedation details, outcome measures, and adverse events. Access will require a data-sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be made available within 6 months after publication of the main results and will remain available for up to 1 year thereafter.
Access Criteria: Qualified researchers affiliated with academic institutions, healthcare organizations, or regulatory agencies will be able to request access to the de-identified individual participant data (IPD), including demographic variables, treatment allocation, sedation response, recovery scores, adverse events, and primary/secondary outcomes. Supporting documents such as the study protocol and statistical analysis plan (SAP) will also be available.
  Access will be granted upon submission and approval of a written data request, which must include a brief research proposal and data use rationale. A data-sharing agreement must be signed prior to access. Data will be shared securely via encrypted files or institutional data-sharing platforms approved by the sponsor institution.
URL: https://www.humanitas-research.com/

REFERENCES:
- See also: Requests should be submitted to: ibd@humanitas.it Subject: REMI-IBD IPD — https://www.humanitas-research.com/
- Available data/document: Study Protocol — https://www.humanitas-research.com/ — Requests should be submitted to: ibd@humanitas.it Subject: REMI-IBD